CLINICAL TRIAL: NCT06220630
Title: The Characteristics, Treatment Patterns and Prognosis of Chinese Male Breast Cancer: A Real-world Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Beijing Medical Award Foundation (Unknown); The Affiliated Cancer Hospital of Xinjiang Medical University (Unknown); Hebei Medical University Fourth Hospital (Other); The Third Affiliated Hospital of Kunming Medical University (Unknown); Sun Yat-sen University (Other); The Affiliated Cancer Hospital of Zhengzhou University (Unknown); The Third Hospital of Nanchang City (Unknown); Beijing 302 Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Fujian Provincial Hospital (Other); First Hospital of China Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First People's Hospital of Foshan (Other); Peking University First Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Jiangmen Central Hospital (Other); The Second Affiliated Hospital, Guangzhou Medical University (Unknown); The First Affiliated Hospital, Zhejiang University (Unknown); Peking University Shenzhen Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Affiliated Sanming First Hospital of Fujian Medical University (Unknown); Jieyang People's Hospital (Other); National Clinical Research Center for Cancer/Cancer Hospital & Shenzhen Hospital (Unknown); Shantou Central Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Lianjiang Pepole's Hospital, Lianjiang (Unknown); Guangdong Women and Children Hospital (Other); Zhanjiang Central Hospital (Unknown); Zhuhai Hospital of Integrated Traditional Chinese and Western Medicine (Unknown)
Responsible Party: Principal Investigator, Ying Lin, MD, PhD, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 2021[516]
Record Dates: First submitted 2024-01-13; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese: About 1,200 Chinese male breast cancer cases are anticipated to collected retrospectively. The clinicopathological characteristics, treatment and survival information are retrospectively collected.
  Interventions: Other: Breast cancer

INTERVENTIONS:
Other: Breast cancer — Male patients who were microscopically diagnosed as primary breast cancer.

SUMMARY:
The goal of this observational study is to investigate the features in Chinese male breast cancer (MBC) patients. The main question it aims to answer is:

* The characteristics, treatment patterns and prognosis of Chinese MBC patients. The clinicopathological characteristics, treatment information and follow-up data of participants will be extracted from a Chinese national database (Chinese Society of Clinical Oncology Breast Cancer database) and other involved Chinese centers.

Researchers will investigate the features, survival associated factors and other relevant factors of this population.

DETAILED DESCRIPTION:
The goal of this observational study is to investigate the features in Chinese male breast cancer (MBC) patients. The main question it aims to answer is:

* The characteristics, treatment patterns and prognosis of Chinese MBC patients. The clinicopathological characteristics, treatment information and follow-up data of participants will be extracted from a Chinese national database (Chinese Society of Clinical Oncology Breast Cancer database) and other involved Chinese centers.

Researchers will investigate the features, survival associated factors and other relevant factors of this population.

The collected variables included: survival time, survival status, year of diagnosis, age, stage, molecular subtype statuses, histology, grade, and surgery, radiotherapy and systemic therapies utilization.

ELIGIBILITY:
Inclusion Criteria:

* Biological sex is male;
* Microscopically diagnosed as primary breast cancer.

Exclusion Criteria:

* Presence of skin-origin malignancy on the breast.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible cases were collected from a Chinese national database (Chinese Society of Clinical Oncology Breast Cancer database) and other involved centers.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the time of diagnosis to August 1, 2024 (anticipated).
  The duration between the date of the first pathologic diagnosis and death from any cause or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lin, MD, PhD, Principal Investigator — 1st affiliated hospital of Sun Yat-sen university
Locations (1):
- First affiliated hospital of Sun Yat-sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
A part of Chinese data that support the findings of this study are available from Chinese Society of Clinical Oncology Breast Cancer Database but restrictions apply to the availability of these data, which were used under license for the current study, and so are not publicly available. Chinese data are however available from the corresponding author upon reasonable request and with permission of Chinese Society of Clinical Oncology Breast Cancer Database.